CLINICAL TRIAL: NCT01532856
Title: Iberoamerican Phase III International Study, Open, Multicenter, Randomized, Comparative of Thalidomide / Cyclophosphamide / Dexamethasone Versus Thalidomide / Dexamethasone Versus Thalidomide / Melphalan / Prednisone as Induction Therapy Followed by Maintenance Therapy With Thalidomide + Prednisone Versus Thalidomide Alone in Patients With Symptomatic Newly Diagnosed Multiple Myeloma Over 65years.
Brief Title: Iberoamerican Protocol With Thalidomide in Patients With Symptomatic Newly Diagnosed Multiple Myeloma Over 65 Years
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo de Estudos Multicentricos em Onco-Hematologia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBRAM0002
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; thalidomide; comparative; elderly
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Cyclophosphamide; Dexamethasone; Melphalan; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A induction therapy (Active Comparator): Thalidomide + Cyclophosphamide + Dexamethasone
  Interventions: Drug: Thalidomide, Cyclophosphamide, Dexamethasone
- Group B induction therapy (Active Comparator): thalidomide + dexamethasone
  Interventions: Drug: Thalidomide, Dexamethasone
- Group C induction therapy (Active Comparator): thalidomide + melphalan + prednisone
  Interventions: Drug: Thalidomide, Melphalan, Prednisone

INTERVENTIONS:
Drug: Thalidomide, Cyclophosphamide, Dexamethasone — Thalidomide - 200mg per day, orally, during 9 cycles of 28 days each cycle Cyclophosphamide - 50mg per day, orally, during 9 cycles of 28 days each cycle Dexamethasone - 40mg orally(two pulses the first two cycles in days 1-4 and 15-18 and then a single pulse in each other cycle) during 9 cycles of 28 days.
  Arms: Group A induction therapy
Drug: Thalidomide, Dexamethasone — Thalidomide - 200mg per day, orally, during 9 cycles of 28 days each cycle Dexamethasone - 40mg orally, in three pulses (days 1 to 4, 9 to 12 and 17 20) odd cycles and a single pulse treatment in pairs cycles, during 9 cycles of 28 days each cycle
  Arms: Group B induction therapy
Drug: Thalidomide, Melphalan, Prednisone — thalidomide - 200mg per day, orally, during 9 cycles of 28 days each cycle; melphalan - 4 mg/m2, days 1-7, orally, during 9 cycles of 28 days each cycle; prednisone - 40 mg/m2, days 1-7, orally, during 9 cycles of 28 days each cycle
  Arms: Group C induction therapy

SUMMARY:
This protocol is an international, multicenter, comparative, open and randomized study designed to compare the safety and efficacy (in terms of response rate) from three induction chemotherapy schemes -Thalidomide/Cyclophosphamide/Dexamethasone versus Thalidomide/Dexamethasone versus Thalidomide/Melphalan/Prednisone. Finally, this study is also designed to compare the safety and efficacy (in terms of duration of response) of two maintenance chemotherapy regimens - Thalidomide/Prednisone versus Thalidomide. Each treatment arm will include 100 patients and assessments and scheduled visits will be conducted in three periods: Pre-treatment, treatment and monitoring. Security will be evaluated by monitoring all adverse events, physical examination, vital signs and biochemical studies. Response to treatment will be evaluated according to the EBMT21 criteria and will be assessed on day 1 of each cycle of induction, at the end of nine cycles of induction therapy and monthly during the first year of maintenance therapy and every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* > 65 years old and non candidate for autologous stem cell transplant
* Patient must be newly diagnosed with Multiple Myeloma according to establish criteria symptoms. Steroid pulses administration are allowed for any required emergency prior to starting induction therapy or bisphosphonates administration
* Patient must have measurable disease, defined as follows: for secretory multiple myeloma, measurable disease is defined by the presence of measurable monoclonal component in serum or in urine excretion if light chain is greater than or equal to 200 mg/24 hours(Annex 5)
* Measured ECOG < 2 state level.
* The patient must have a life expectancy greater than 3 months.
* Adequate laboratory values prior to induction treatment initiation, defined as follow:

  1. Platelet count ≥ 50000/mm3, hemoglobin ≥ 8 g / dl and absolute neutrophil count ≥ 1000/mm3. Lower values are permitted if they are due to BM infiltration.
  2. Corrected serum calcium ≤ 14mg/dl.
  3. Aspartate transaminase (AST): ≤ 2.5 x normal upper limit.
  4. Alanine transaminase (ALT):): ≤ 2.5 x normal upper limit.
  5. Total bilirubin: ≤ 1.5 x normal upper limit.
  6. Serum creatinine ≤ 2 mg / dl.
* Men (including vasectomy done) must use barrier contraception (latex condoms) when having sex with women of potential childbearing, and for at least four weeks after thalidomide last dose.

Exclusion Criteria:

* Non-secretory MM.
* Previous treatment for multiple myeloma with the exception of steroid pulses for any emergency that requires treatment before beginning the induction, administration of bisphosphonates or radiation therapy.
* Basal peripheral neuropathy higher than grade 2 within 14 days of inclusion.
* Known thalidomide hypersensitivity.
* Use of any investigational agent within 30 days prior to their inclusion.
* Known human immunodeficiency virus(HIV) infection, detectable surface antigen of hepatitis B or active infection by the hepatitis C viruses
* Myocardial infarction within 6 months prior to inclusion or heart functional class III or IV according to New York Heart Association (NYHA) heart failure, angina, uncontrolled ventricular arrhythmias or acute ischemia detected by electrocardiogram or conduction system abnormalities.
* Participation in another clinical trial or receiving any investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2007-01; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Response rate | 36 months
  Response rate is evaluated between the 3 treatment arms
Duration of response | 36 months
  Duration of response was defined as the time to the first evidence of laboratorisl progreesion.

SECONDARY OUTCOMES:
overall survival | 36 months
  Overall survival (OS) was defined as the interval from randomization to death or the last follow-up for surviving patients.
event-free survival | 36 months
  Event-free survival was defined as the interval from randomization to any event (death or descontinuation due to protocol violation or non-acceptable toxicities)
progression free-survival | 36 months
  Progression free-survival was defined as the time between randomization and any documentation of relapse, progression, or death by any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Vania Hungria, PhD MD, Principal Investigator — Santa Casa de Misericordia de São Paulo
Locations (3):
- Brazil (3):
  - Hospital Universitário Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro
  - Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo